CLINICAL TRIAL: NCT04535908
Title: Clinical Study to Evaluate Hypofractionated Radiotherapy in Prostate Cancer Patients Aged 75 Years or Older.
Brief Title: Hypofractionated Radiotherapy in Prostate Cancer Patients Aged 75 Years or Older.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Treatment standard has changed.
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1091/2020
Record Dates: First submitted 2020-08-25; First posted 2020-09-02 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Prostate Cancer; Radiotherapy Side Effect
Keywords: Hypofractionated radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms; Radiation Injuries | interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypofractionated radiotherapy (Experimental)
  Interventions: Radiation: Hypofractionated radiotherapy

INTERVENTIONS:
Radiation: Hypofractionated radiotherapy — Hypofractionated radiotherapy in prostate cancer patients

SUMMARY:
The majority of all new prostate cancer cases are diagnosed in men aged > 70 years, with the highest incidence in men aged > 90 years. Management options for localized prostate cancer include active surveillance in patients with low-risk disease, radical prostatectomy or external beam radiation therapy.

In previous studies, hypofractionated prostate cancer irradiation regimens have been shown to represent a highly effective treatment option for prostate cancer. However, patients aged 75 years or older were underrepresented in most trials resulting in the lack of a robust evidence base.

The proposed study will evaluate radiation-induced toxicity as well as outcome after hypofractionated external beam radiotherapy in prostate cancer patients aged 75 years or older.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed prostate cancer adenocarcinoma
* definitive radiotherapy for curative intent
* low or intermediate risk prostate cancer
* patient age ≥ 75 years
* given informed consent

Exclusion Criteria:

* chronic inflammatory bowel disease
* high risk prostate cancer
* lymph node or distant metastases
* unable to give informed consent

Min Age: 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Acute radiation - induced toxicity | Measurement at the last 1 day of radiotherapy
  Toxicity score using Common Terminology for Adverse Events (CTCAE)
Acute radiation - induced toxicity | Measurement 3 months after completion of radiotherapy
  Toxicity score using Common Terminology for Adverse Events (CTCAE)

SECONDARY OUTCOMES:
Overall survival | At 1, 2, 3 , 4, 5 years after completion of radiotherapy
  Analysis of survival
Recurrence (biochemical) | At 1, 2, 3 , 4, 5 years after completion of radiotherapy
  Assessed by measurement of prostate specific antigen (PSA)
Recurrence (local) | At 1, 2, 3 , 4, 5 years after completion of radiotherapy
  Assessed by magnetic resonance imaging (MRI), positron emission tomography (optional)

CONTACTS AND LOCATIONS:
Overall Officials: Tanja Langsenlehner, MD, Principal Investigator — Medical University of Graz, Dept. of Therapeutic Radiology and Oncology
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dearnaley D, Syndikus I, Mossop H, Khoo V, Birtle A, Bloomfield D, Graham J, Kirkbride P, Logue J, Malik Z, Money-Kyrle J, O'Sullivan JM, Panades M, Parker C, Patterson H, Scrase C, Staffurth J, Stockdale A, Tremlett J, Bidmead M, Mayles H, Naismith O, South C, Gao A, Cruickshank C, Hassan S, Pugh J, Griffin C, Hall E; CHHiP Investigators. Conventional versus hypofractionated high-dose intensity-modulated radiotherapy for prostate cancer: 5-year outcomes of the randomised, non-inferiority, phase 3 CHHiP trial. Lancet Oncol. 2016 Aug;17(8):1047-1060. doi: 10.1016/S1470-2045(16)30102-4. Epub 2016 Jun 20. PMID 27339115